CLINICAL TRIAL: NCT05130710
Title: The Impact of COVID-19 Pandemic on Clinical Presentation and Staging of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IR.TUMS.IKHC.REC.1399.414
Record Dates: First submitted 2021-11-19; First posted 2021-11-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Gastric Cancer; COVID-19 Pandemic; Peritoneal Metastases
MeSH Terms: conditions — Stomach Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — in time of performing staging laparoscopy if any suspicious tissue for being malignant was encounter biopsied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: 26 patients with gastric cancer wo were referred to our center between February 25th to December 25th of 2020.
  Interventions: Procedure: staging laparoscopy
- control: 54 patients with gastric cancer wo were referred to our center between February 25th to December 25th of 2019.
  Interventions: Procedure: staging laparoscopy

INTERVENTIONS:
Procedure: staging laparoscopy — All patients of both groups underwent staging laparoscopy by the same two attending onco-surgeon, using the same technique and the same laparoscopic device. Under general anesthesia and in supine position SL was performed. A 10 mm optic laparoscopic port was inserted via the midline incision below the umbilicus using Hasson technique. All four quadrants of the abdomen as well as pelvis were inspected during laparoscopy and biopsy was taken from any suspicious lesion through insertion of 5mm port. All specimens underwent cytological evaluation by two independent pathologists. The presence of any malignant cells, regardless of the number, confirmed the positive cytology. In the event of discordant reports between two pathologists, specimens were sent for the third review by a pathologist who was blinded to the previous results. Laparoscopic evaluation was considered positive as if adjacent organ involvement, omental involvement or peritoneal seeding were seen.

SUMMARY:
This was a retrospective case-control study designed and conducted under the approval of the ethic committee of Tehran University of Medical Sciences. All patients with gastric cancer referring to Cancer Institute, Tehran University of Medical Sciences, Tehran, Iran, during February 25th and December 25th 2020, were enrolled to the study.

DETAILED DESCRIPTION:
This was a retrospective case-control study designed and conducted under the approval of the ethic committee of Tehran University of Medical Sciences. All patients with gastric cancer referring to Cancer Institute, Tehran University of Medical Sciences, Tehran, Iran, during February 25th and December 25th 2020, were enrolled to the study. February 25th was the day Ministry of Health and Medical Education announced COVID-19 as a national disaster and set restrictive rules of social distancing. The control group consisted of the gastric cancer patients whom referred to Cancer Institute during February 25th and December 25th of 2019. So the investigators compared two groups of gastric cancer patients one in the era of COVID-19 pandemic and other group from previous year when there was no COVID-19.

Cancer Institute as the pioneer of cancer management in Iran set institutional regulation for hospitalization of cancer patients during COVID-19 pandemic with the primary goal of delivering the best available treatment as timely as possible. In order to achieve this, each patient regardless of cancer type must had proceeded these steps before elective hospitalization and during preoperative, operation and postoperative days:

1. Prior to hospitalization, patients were referred to infectious disease clinic, where they were visited by attending infectious disease specialists who had fellowship in infectious disease of immunocompromised and transplanted patients. Every patient monitored for COVID-19 sign and symptoms and those with high susceptibility were examined utilizing spiral chest computed tomography scan (SCCT) and polymerase chain reaction (PCR) for SARS-CoV-2. If a patient had positive result of either SCCT or PCR, he/she was managed either in outpatient or inpatient setting for COVID-19 treatment based on national protocol and subsequent cancer management was postponed. If it was confirmed that patient is eligible for hospitalization and entering operation room, he/she was admitted to surgical oncology ward.
2. During pre-operative days, all patients were hospitalized in single or double bed room, family members were not allowed to accompany except for under legal aged patient and those who need special attention because of the low performance status. All patients were educated about COVID-19 transmission routs and preventive measures and asked to respect social distancing, wear facial mask and wash hands using alcohol- based antiseptic formulas given. Each patient underwent daily monitoring for sign and symptoms of COVID-19, heart rate, blood pressure, temperature and oxygen saturation by commercially available pulse oximetry devices. In case of developing signs and symptoms related to COVID-19 or unexplained temperature > 38°C, oxygen saturation < 93% or > 5 unit drop in oxygen saturation from the baseline, infectious disease consultation was ordered.
3. During operation time, the minimum number of personnel needed to activate a safe operation environment whom were fully equipped with personal preventive clothing including surgical cap, gown, facial mask and shield were present at the theater. The operation theater was well ventilated.
4. During post-operative days, for both intensive care unit and ward patient, daily monitoring of signs and symptoms related to COVID-19 besides unexplained temperature > 38°C, oxygen saturation < 93% or > 5 unit drop in oxygen saturation from the baseline, C-Reactive Protein Level > 40 persistent for 3 days activated infectious disease consultation.

Patients of both case and control group were enrolled to the study as if they gave written consent of participation, had confirmed gastric cancer using esophago-gastro-duodenoscopy and pathologically proven biopsy and spiral thoraco-abdomino-pelvic computed tomography scan prior to surgery. All patients became candidates to undergo staging laparoscopy (SL) in order to investigate local and peritoneal invasion of the tumor based on National Comprehensive Cancer Network guideline for gastric cancer 2020. Patients with following criteria were excluded from the study; radiological evidence of metastatic disease, current or previous history of chemotherapy.

All patients of both groups underwent SL by the same two attending onco-surgeon, using the same technique and the same laparoscopic device. Under general anesthesia and in supine position SL was performed. A 10 mm optic laparoscopic port was inserted via the midline incision below the umbilicus using Hasson technique. All four quadrants of the abdomen as well as pelvis were inspected during laparoscopy and biopsy was taken from any suspicious lesion through insertion of 5mm port. All specimens underwent cytological evaluation by two independent pathologists. The presence of any malignant cells, regardless of the number, confirmed the positive cytology. In the event of discordant reports between two pathologists, specimens were sent for the third review by a pathologist who was blinded to the previous results. Laparoscopic evaluation was considered positive as if adjacent organ involvement, omental involvement or peritoneal seeding were seen.

Data were collected on the following variables: age, gender, tumor location, gastric lesion pathology and clinical stage based on the 8th edition of the American Joint Committee on Cancer tumor-node metastasis staging system for gastric cancer[16].

Categorical variables are shown as number and relative frequency. Also, continuous variables are shown as mean ± SD. Collected data for categorical variables were compared using the chi-squared test. An independent student t-test was used to compare means between the two groups. All analyses were performed by the two-sided method using Statistical Package of Social Science software (SPSS version 22; SPSS, Inc., Chicago, IL), and the p-value of < 0.05 was set as statistically signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

All patients became candidates to undergo staging laparoscopy (SL) in order to investigate local and peritoneal invasion of the tumor based on National Comprehensive Cancer Network guideline for gastric cancer 2020.

Exclusion Criteria:

Patients with following criteria were excluded from the study; radiological evidence of metastatic disease, current or previous history of chemotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with gastric cancer referring to Cancer Institute, Tehran University of Medical Sciences, Tehran, Iran, during February 25th and December 25th 2020, were enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
presence of peritoneal seeding | February 25th and December 25th 2020
  involvement of peritoneal cavity with metastatic gastric cancer.

SECONDARY OUTCOMES:
presence of peri-gastric lymph node involvement | February 25th and December 25th 2020
  involvement of peri-gastric lymph node with metastatic gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer institute, Imam Khomeini Hospital Complex, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
data will be available up on reasonable request from Amirisina Sharifi.M.D.(a.s_sharifi@yahoo.com).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Salari A, Jalaeefar A, Shirkhoda M. What is the best treatment option for head and neck cancers in COVID-19 pandemic? A rapid review. Am J Otolaryngol. 2020 Nov-Dec;41(6):102738. doi: 10.1016/j.amjoto.2020.102738. Epub 2020 Sep 18. PMID 32979663
- [Background] Di Fiore F, Bouche O, Lepage C, Sefrioui D, Gangloff A, Schwarz L, Tuech JJ, Aparicio T, Lecomte T, Boulagnon-Rombi C, Lievre A, Manfredi S, Phelip JM, Michel P; Thesaurus National de Cancerologie Digestive (TNCD); Societe Nationale Francaise de Gastroenterologie (SNFGE); Federation Francophone de Cancerologie Digestive (FFCD); Groupe Cooperateur multidisciplinaire en Oncologie (GERCOR); Federation Nationale des Centres de Lutte Contre le Cancer (UNICANCER); Societe Francaise de Chirurgie Digestive (SFCD); Societe Francaise d'Endoscopie Digestive (SFED); Societe Francaise de Radiotherapie Oncologique (SFRO) and Societe Francaise de Radiologie (SFR); Association Chirurgie Hepato-Biliaire et Transplantation (ACHBT). COVID-19 epidemic: Proposed alternatives in the management of digestive cancers: A French intergroup clinical point of view (SNFGE, FFCD, GERCOR, UNICANCER, SFCD, SFED, SFRO, SFR). Dig Liver Dis. 2020 Jun;52(6):597-603. doi: 10.1016/j.dld.2020.03.031. Epub 2020 May 14. PMID 32418773
- [Background] Johnson BA, Waddimba AC, Ogola GO, Fleshman JW Jr, Preskitt JT. A systematic review and meta-analysis of surgery delays and survival in breast, lung and colon cancers: Implication for surgical triage during the COVID-19 pandemic. Am J Surg. 2021 Aug;222(2):311-318. doi: 10.1016/j.amjsurg.2020.12.015. Epub 2020 Dec 8. PMID 33317814
- [Background] Wu JT, Kwon DH, Glover MJ, Henry S, Wood D, Rubin DL, Koshkin VS, Schapira L, Shah SA. Changes in Cancer Management due to COVID-19 Illness in Patients with Cancer in Northern California. JCO Oncol Pract. 2021 Mar;17(3):e377-e385. doi: 10.1200/OP.20.00790. Epub 2020 Dec 17. PMID 33332170
- [Background] Zaniboni A, Ghidini M, Grossi F, Indini A, Trevisan F, Iaculli A, Dottorini L, Moleri G, Russo A, Vavassori I, Brevi A, Rausa E, Boni L, Dondossola D, Valeri N, Ghidini A, Tomasello G, Petrelli F. A Review of Clinical Practice Guidelines and Treatment Recommendations for Cancer Care in the COVID-19 Pandemic. Cancers (Basel). 2020 Aug 29;12(9):2452. doi: 10.3390/cancers12092452. PMID 32872421
- [Background] Chan JW, Lee VHF. Will the COVID Pandemic Lead to Uncounted Cancer Deaths in the Future? Int J Radiat Oncol Biol Phys. 2020 Oct 1;108(2):351-352. doi: 10.1016/j.ijrobp.2020.07.003. No abstract available. PMID 32890510
- [Background] Vanni G, Tazzioli G, Pellicciaro M, Materazzo M, Paolo O, Cattadori F, Combi F, Papi S, Pistolese CA, Cotesta M, Santori F, Caspi J, Chiaravalloti A, Muscoli S, Lombardo V, Grasso A, Caggiati L, Raselli R, Palli D, Altomare V, D'Angelillo RM, Palombi L, Buonomo OC. Delay in Breast Cancer Treatments During the First COVID-19 Lockdown. A Multicentric Analysis of 432 Patients. Anticancer Res. 2020 Dec;40(12):7119-7125. doi: 10.21873/anticanres.14741. Epub 2020 Dec 7. PMID 33288611
- [Background] Gundavda MK, Gundavda KK. Cancer or COVID-19? A Review of Guidelines for Safe Cancer Care in the Wake of the Pandemic. SN Compr Clin Med. 2020;2(12):2691-2701. doi: 10.1007/s42399-020-00632-2. Epub 2020 Nov 21. PMID 33251481
- [Background] Arpino G, De Angelis C, De Placido P, Pietroluongo E, Formisano L, Bianco R, Fiore G, Montella E, Forestieri V, Lauria R, Cardalesi C, Vozzella EA, Iervolino A, Giuliano M, De Placido S. Optimising triage procedures for patients with cancer needing active anticancer treatment in the COVID-19 era. ESMO Open. 2020 Sep;5(5):e000885. doi: 10.1136/esmoopen-2020-000885. PMID 32958531